CLINICAL TRIAL: NCT00000787
Title: Heterosexual HIV Transmission Study (HATS). Prospective Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: HATS PROSPECTIVE
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: HIV Infections
Keywords: Sex Behavior
MeSH Terms: conditions — HIV Infections; Sexual Behavior | interventions — Lead

INTERVENTIONS:
Behavioral: Pre- and post-test counseling

SUMMARY:
PRIMARY: To identify factors associated with risk of HIV infection through heterosexual activity among urban, inner-city women.

SECONDARY: To identify correlates of high-risk behaviors in order to provide a basis for future intervention studies.

DETAILED DESCRIPTION:
At baseline and at 6-month intervals, participants are interviewed about their sexual behavior, drug and alcohol-related behaviors, and recent medical history, and are given a psychosocial assessment. They also undergo a physical exam, including pelvic exam and colposcopy, and have blood and urine specimens collected for HIV testing, drug screening, and STD evaluation. Additionally, participants are given pre- and post-test counseling and education, including information about social services. They are provided with basic gynecological care and either treatment or referral for medical problems.

ELIGIBILITY:
Participants must meet the following criteria:

* HIV-negative, sexually active women living in social and sexual proximity to men at high risk for acquiring HIV infection.
* Able to speak English, Spanish, or Creole.
* Living in the geographic area surrounding Kings County Hospital in Brooklyn, New York. (Hospital-based and community-based recruitment sites will be utilized.)

Personal history of parenteral drug use by self-report or urine test. Heterosexual contact with men at high risk for HIV infection.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York, United States

REFERENCES:
- [Background] Skurnick J, Bromberg J, Cordell J, Foley M, Wang W, Louria D. Change in couples' sexual activity after knowledge of HIV discordance: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(2):C273 (abstract no PoC 4170)
- [Background] Skurnick J, Bromberg J, Grijalva K, Cordell J, Louria D, Monto A, Weiss S. Behavior changes in heterosexual couples discordant for HIV: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1991 Jun 16-21;7(2):319 (abstract no WC3094)
- [Background] Padian N, Bromberg J, O'Brien T, Vranizan K, Cordell J, Louria D, Van-Devanter N, Landesman S. Smoking and bleeding from trauma during sex: risks for heterosexual transmission of HIV. The HATS/CDC Research Group. Int Conf AIDS. 1993 Jun 6-11;9(2):648 (abstract no PO-C02-2588)
- [Background] Wan J, Bromberg J, Cornell RG, Skurnick J, Cordell J, Vermund S. Generalized additive models for paired covariates in an HIV discordant couples study: a report from The Heterosexual HIV Transmission Study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(3):193 (abstract no PuC 8243)
- [Background] Bromberg J, Wan J, Cornell RG, Grijalva K, Cordell J, Kelly P, Landesman S. Entry criteria bias in studies of high-risk individuals: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(2):C371 (abstract no PoC 4773)
- [Background] Bromberg J, Maher J, Wang W, Grijalva K, Cordell J. Within couple disagreement on condom use: a report from the heterosexual HIV transmission study (HATS/CDC). Int Conf AIDS. 1993 Jun 6-11;9(2):774 (abstract no PO-C33-3345)
- [Background] Sogolow ED, Des Jarlais D, Landesman SH, Kelly P, Sampson-Lee G, Cordell J, Cornell R. The experience of participating in a cohort study of HIV transmission: a report from The Heterosexual HIV Transmission Study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(3):189 (abstract no PuC 8216)
- [Background] Cornell RG, Bromberg J, Grijalva K, Kelly P, Cordell J. Effects of changing recruitment patterns on risk factor estimates: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(2):C324 (abstract no PoC 4477)
- [Background] Strug D, Des Jarlais D, Sogolow E, Handte J, Bromberg J, Cornell R, Cordell J, Landesman S. Types of sexual partner relationships and condom use among women in Brooklyn: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1991 Jun 16-21;7(2):324 (abstract no WC3112)